CLINICAL TRIAL: NCT00965913
Title: Study on the Cumulative Skin Irritation Potential of a Newly Developed 15 mg Nicotine Transdermal Therapeutic System. A Double Blind, Randomized, Repeat Patch Test, Single Center Study in 42 Healthy Male and Female Subjects
Brief Title: Cumulative Skin Irritation Potential of a New 15 mg Nicotine Patch
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: A6431082; 2005-001044-23 (EudraCT Number); 012/05-03.NSI (Other: CRO)
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Three Interventions on Lower Back (Experimental): Three treatments were applied on the lower back, according to treatment sequence, daily for 21 days
  Interventions: Drug: Nicotine Patch; Drug: Nicotine Patch Comparator; Drug: Placebo Patch

INTERVENTIONS:
Drug: Nicotine Patch — 15 mg nicotine patch applied on the lower back, according to treatment sequence, daily for 21 days
  Other Names: Experimental Nicotine Patch
Drug: Nicotine Patch Comparator — 15 mg nicotine patch applied on the lower back, according to treatment sequence, daily for 21 days
  Other Names: Active Comparator Nicotine Patch
Drug: Placebo Patch — Placebo patch applied on the lower back, according to treatment sequence, daily for 21 days
  Other Names: Placebo Patch Comparator

SUMMARY:
An investigation on the cumulative skin irritation potential of a newly developed 15 mg nicotine patch. Evaluation of skin irritation of a newly developed 15 mg nicotine transdermal patch.

DETAILED DESCRIPTION:
Study on the cumulative skin irritation potential of a newly developed 15 mg nicotine transdermal therapeutic system. A double blind, randomized, repeat patch test, single center study in 42 healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 and 65 years
* Heavy smokers (more than 10 cigarettes per day)
* Having had no febrile or infectious illness for at least seven days prior to the first administration of the investigational product.
* Women practicing one or a combination of the following methods of birth control: hormonal contraceptives, condoms, sponge, foams, jelly, diaphragm, or intrauterine device or women who are surgically sterilized.
* Subjects having normal skin without excessive hair growth on tested areas.
* Evidence of a personally signed and dated informed consent document indicating that the subjects has been informed of all pertinent aspects of the trial.
* Subjects who are willing to comply with scheduled visits, treatment plan and other trial procedures.

Exclusion Criteria:

* Any visible skin disorder or abnormal skin pigmentation which, in the opinion of the investigator, would interfere with the outcome of the trial
* Dermatologic disease that might interfere with the evaluation of the test site reaction
* History of chronic, dermatological, medical, or physical conditions which would, in the opinion of the investigator, preclude topical application of the test products and/or influence the outcome of the test (in particular, any immunosuppressive condition)
* Clinically relevant abnormal findings on the physical examination
* A baseline score in skin reaction assessments other than "0" on the areas to be patched
* Pregnant (verified by beta-hCG-test in urine) and/or nursing women
* Demonstrating any active physical disease, acute or chronic
* Any suspicion, history or evidence of alcohol or drug abuse
* Any history of drug hypersensitivity, asthma, urticaria or other severe allergic diathesis as well as current hay fever
* Any current or past history of chronic or recurrent metabolic, renal, hepatic, pulmonary, gastrointestinal, neurological, endocrinological, immunological, psychiatric or cardiovascular disease, myopathies, epileptic seizures and bleeding tendency
* Recent myocardial infarct (within the last 3 months), unstable or deteriorating angina pectoris, coronary artery vasospasm (Prinzmetal's angina), serious cardiac arrythmias and acute stroke
* Use of any medication within 4 weeks prior to the first treatment or during the trial, which in the opinion of the investigator may influence the trial results or the safety of the subjects
* Subjects having used nicotine products other than cigarettes within the 3 months preceding the trial or within 10 times the respective elimination half-life, whichever is longer
* Subjects who cannot avoid, throughout the duration of the trial, any swimming, any washing of the back and sauna or any intense physical activity that might result in excessive sweating
* Known sensitivity to adhesive tape
* Known sensitivity to any component of the test products
* History of irritation to topically applied products
* Fissure or injury of the skin at the test area
* Participation in the treatment phase of a clinical trial within 30 days prior to the treatment phase of this trial or within 10 times the respective elimination half-life of the investigational drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-05; Primary Completion 2005-05 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Cumulative Irritation Score (CIS10) | @24 hours post- application for 21 days

SECONDARY OUTCOMES:
Cumulative Individual Irritation Score (CIIS) | @24 hours post- application for 21 days
Frequency Indices (FI) of irritation score | @24 hours post- application for 21 days
Time to irritation reaction | @24 hours post- application for 21 days
Patch adhesion score | directly before patch removal
Tolerability | at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — Mc Neil AB
Locations (1):
- IKP, Mannheim, Germany